CLINICAL TRIAL: NCT00726596
Title: NJ 1808: Autophagic Cell Death With Hydroxychloroquine in Patients With Hormone-Dependent Prostate-Specific Antigen Progression After Local Therapy For Prostate Cancer.
Brief Title: Hydroxychloroquine in Treating Patients With Rising PSA Levels After Local Therapy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Biren Saraiya, MD, Assistant Professor of Medicine Medical Oncology, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0220080115; P30CA072720 (NIH); 0220080115 (Other: IRB); NCI-2012-00528 (Other: NCI #); 080803 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2008-07-31; First posted 2008-08-01 (Estimated); Results first posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer; Prostate-Specific Antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxychloroquine (Experimental): Hydroxychloroquine - 400 mg (cohort A) Hydroxychloroquine - 600 mg (cohort B)
  Interventions: Drug: hydroxychloroquine

INTERVENTIONS:
Drug: hydroxychloroquine — Hydroxychloroquine will be taken at a dose of 200 mg twice per day in the first 27 patients (cohort A). Once cohort A completed, the dose of hydroxychloroquine will then be increased to 600mg per day (200mg three times per day)(cohort B).

SUMMARY:
This phase II trial studies how well hydroxychloroquine works in treating patients with previously treated prostate cancer. Autophagy destroys proteins and other substances in cells and may be used by prostate cancer cells to survive. Hydroxychloroquine, which blocks autophagy, may slow the growth of and possibly kill prostate cancer cells.

ELIGIBILITY:
Inclusion Criteria

* Histologically proven stage D0 prostate cancer (i.e., tumor originally diagnosed as being limited to the prostate) or D1 prostate cancer (metastatic to regional lymph nodes) and have a rising PSA value after definitive local therapy.
* Must have undergone local treatment via prostatectomy or radiation therapy.
* Must have PSA progression after local treatment:

  1. PSA values for patients after surgery must be > 0.2 ng/mL, determined by two measurements, at least 1 month apart and at least 6 months after prostatectomy
  2. PSA values for patients after radiation must be ≥ 2.0 ng/ml greater than the nadir achieved after radiation, determined by two measurements at 1 month apart and at least 6 months after the radiation treatment is completed. (Patients who received adjuvant or salvage radiation after prostatectomy must have PSA of >0.2)
  3. The first two PSA values (in 5.1.3a and 5.1.3b), along with a third (study baseline) value must all be rising (i.e., there must be an overall rising trajectory, such that the third value cannot be lower than the first value).
* Baseline bone scan and CT abdomen/pelvis demonstrating no metastatic disease.
* Age ≥ 18 years
* Estimated life expectancy of at least 6 months.
* ECOG performance status < 2. (see Appendix B)
* A WBC > 3500/μl, ANC >1500/μl, hemoglobin > 10 g/dl, and platelet count >100,000/μl are required.
* Adequate renal function (serum creatinine < 1.5 mg/dL or creatinine clearance > 50 ml/min).
* Total bilirubin must be within 1.5X the normal institutional limits. If total bilirubin is outside the normal institutional limits, assess direct bilirubin. The direct bilirubin must be within normal parameters. Transaminases (SGOT and/or SGPT) must be less than 2.5X the institutional upper limit of normal.
* Documented ophthalmic exam within the last twelve months demonstrating no evidence of retinopathy. Patients with retinal changes will be considered for enrollment with written clearance from a board certified ophthalmologist.
* Must have a serum total testosterone level ≥150 ng/dL at the time of enrollment within 4 weeks prior to randomization.
* Must sign informed consent.

Exclusion Criteria

* Serious concomitant systemic disorder that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Must be off ADT in the neoadjuvant, adjuvant and/or salvage setting for at least 3 months and have a testosterone level > 150 ng/dl.
* Second primary malignancy except most situ carcinoma (e.g. adequately treated non-melanomatous carcinoma of the skin) or other malignancy treated at least 5 years previously with no evidence of recurrence.
* Rheumatoid arthritis or systemic lupus erythematosus treatment.
* Psoriasis.
* Receiving any disease-modifying anti-rheumatic drug (DMARD).
* Active clinically significant infection requiring antibiotics.
* G6PD deficiency.
* Taking other commercially available medications which may theoretically either stimulate or inhibit autophagy, which are calcitriol and chloroquine.
* Taking medications which may lead to interactions with hydroxychloroquine, including penicillamine, telbivudine, botulinum toxin, digoxin, and propafenone.
* Must not have visual field changes from prior 4-aminoquinoline compound use.
* Must not be taking hydroxychloroquine for treatment or prophylaxis of malaria.
* History of hypersensitivity to 4-aminoquinoline compound.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-08; Primary Completion 2014-02 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biren Saraiya, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (5):
- United States (5):
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Cooper University Hospital Cancer Institute, Voorhees Township, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey Oncology Group. The study was open to accrual on 08/05/2008 and closed to accrual to 04/10/2013
Pre-assignment Details: We are reporting results on 64 eligible patients. 14 patients were deemed ineligible.
Groups:
- Cohort A. Hydroxychloroquine (200mg Bid): Hydroxychloroquine - 400 mg (cohort A)
  Hydroxychloroquine will be taken at a dose of 200 mg twice per day in the first 27 patients (cohort A).
- Cohort B. Hydroxychloroquine (200mg Tid): Hydroxychloroquine - 600 mg (cohort B)
  Once cohort A is completed, the dose of hydroxychloroquine will then be increased to 600mg per day (200mg three times per day)(cohort B).
Period: Overall Study
Arm/Group | Cohort A. Hydroxychloroquine (200mg Bid) | Cohort B. Hydroxychloroquine (200mg Tid)
Started | 36 | 28
Completed | 31 | 24
Not Completed | 5 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A. Hydroxychloroquine (200mg Bid) | Cohort B. Hydroxychloroquine (200mg Tid) | Total
Number analyzed (Participants) | 36 | 28 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 31 | 19 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 28 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 36 | 28 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 31 | 24 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 28 | 64

OUTCOME MEASURES:

1. Primary Outcome: Prostate-specific Antigen (PSA) Response
Description: PSA response will be defined as a change in slope of at least 25%, when log (PSA) is plotted vs. time
Time Frame: 6 years
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A. Hydroxychloroquine (200mg Bid) | Cohort B. Hydroxychloroquine (200mg Tid)
Number analyzed (Participants) | 30 | 22
percentage of participants | 48 | 48
Statistical Analysis 1: Comparison: Cohort A. Hydroxychloroquine (200mg Bid) vs Cohort B. Hydroxychloroquine (200mg Tid); Test type: Superiority; p = .6789, t-test, 1 sided

2. Secondary Outcome: Effect on Peripheral Blood Mononuclear Cell (PBMC) LC3 Expression by the Use of Hydroxychloroquine
Description: A change of at least 25% from baseline will be considered to be a significant response
Time Frame: 6 years
Population: Data was not collected and the outcome measure was not analyzed.
Arm/Group | Cohort A. Hydroxychloroquine (200mg Bid) | Cohort B. Hydroxychloroquine (200mg Tid)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Effect on PBMC Autophagic Vesicle Formation by the Use of Hydroxychloroquine
Time Frame: 6 years
Population: Data was not collected and the outcome measure was not analyzed.
Arm/Group | Cohort A. Hydroxychloroquine (200mg Bid) | Cohort B. Hydroxychloroquine (200mg Tid)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Expression of Beclin-1 in a Population of Patients Having Undergone Local Treatment With Prostatectomy
Time Frame: 6 years
Population: Data was not collected and the outcome measure was not analyzed.
Arm/Group | Cohort A. Hydroxychloroquine (200mg Bid) | Cohort B. Hydroxychloroquine (200mg Tid)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Feasibility and Safety of Administering Hydroxychloroquine in This Population of Patients. Rate of Adverse Events
Description: Rate of adverse events were captured utilizing the CTCAE version3.0.
Time Frame: 6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A. Hydroxychloroquine (200mg Bid) | Cohort B. Hydroxychloroquine (200mg Tid)
Number analyzed (Participants) | 30 | 22
Participants | 30 | 22

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 170 days per patient.
Arm/Group | Cohort A. Hydroxychloroquine (200mg Bid) | Cohort B. Hydroxychloroquine (200mg Tid)
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/28
Other Adverse Events (participants affected / at risk) | 20/36 | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A. Hydroxychloroquine (200mg Bid) (N=36) | Cohort B. Hydroxychloroquine (200mg Tid) (N=28)
Pain (Renal and urinary disorders) | 1 (1) | 0 (0) — Right flank
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A. Hydroxychloroquine (200mg Bid) (N=36) | Cohort B. Hydroxychloroquine (200mg Tid) (N=28)
Diarrhea (Gastrointestinal disorders) | 20 (20) | 23 (23)
Nausea (Gastrointestinal disorders) | 20 (20) | 7 (7)
Fatigue (General disorders) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Vision - blurred vision (Eye disorders) | 3 (3) | 2 (2)
Allergic rhinitis (Immune system disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 3 (3) | 2 (2) — Headache
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Insomnia (General disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (5)
Pain (General disorders) | 1 (1) | 2 (2) — Back pain
Creatinine (Investigations) | 0 (0) | 3 (3)
Glucose, serum high (Investigations) | 0 (0) | 4 (4)
Hyperkalemia (Investigations) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Research correlatives were not analyzed because the study was unfunded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes